CLINICAL TRIAL: NCT06009120
Title: Impact of Psychosexual Development Theory-Based Breastfeeding Education on Infant Feeding Attitudes and Knowledge of Primiparous Mothers: A Randomized Controlled Study
Brief Title: Psychosexual Development Theory-Based Breastfeeding Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching Assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Eyşan Hanzade Savaş
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding; Psychosocial Development; Nursing Caries
MeSH Terms: conditions — Breast Feeding | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Patients who met the sample selection criteria were randomly divided into two groups, an intervention (education) group and a CG, using a computer-based program (www.random.org). The assignment to the intervention and CG was performed by an independent statistician. Thus, by implementing randomized allocation and concealing the randomization, selection bias was controlled. In the study, participant blinding was carried out, but researcher blinding was not possible due to the researcher's awareness of the intervention being administered. In a 1:1 ratio, the women were separated into intervention and CGs (Figure 1).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention (education) group:
  In addition to the standard discharge education, mothers in this group received breastfeeding education.
  Interventions: Other: Education
- Control (No Intervention): Control group: In this group, first of all, mothers were informed about the study within the first day after birth, and informed consent forms were signed by those who voluntarily agreed to participate. In addition, "Personal Information Form", "IOWA Infant Feeding Attitude Scale" and "Psychosexual Theory and Breastfeeding Information Scale" were applied to these mothers on the first day. Then, as the routine care of the institution, the standard discharge education program on the third day was applied by the institution nurse. After this education, "IOWA Infant Feeding Attitude Scale" and "Psychosexual Theory and Breastfeeding Knowledge Form" were re-administered to mothers as a post-test. No additional intervention was applied other than standard care education. During the 5 days following discharge, mothers were interviewed by phone and "Breastfeeding Form'' applied.

INTERVENTIONS:
Other: Education — The education program emphasized the characteristics of the oral stage, positive traits that can be acquired when the baby's needs are met during this stage, negative traits that may develop in the baby when their needs are not met, and the relationship between the oral stage and breastfeeding.
  Arms: Intervention

SUMMARY:
Breastfeeding education based on the theory of psychosexual development is important as it addresses the social and psychological significance of childhood and the impact of early childhood experiences on later social anxieties and psychosexual well-being. However, no theory-based breastfeeding education given to the mothers was found in the literature. Therefore, the study aimed to investigate the effect of breastfeeding education on infant feeding attitudes and knowledge of primiparous mothers, in line with the theory of psychosocial development.

DETAILED DESCRIPTION:
Breastfeeding is known to play a health-enhancing and disease-preventive role for both the mother and the baby. While it is recognized to reduce postpartum blood loss in mothers and provide protection against conditions like depression, Type 2 diabetes, hypertension, and breast & ovarian cancer; for infants, it is noted that breastfeeding offers protection against many infectious diseases due to the antibodies it, reduces sudden infant deaths and decreases mortality under the age of five [6]. However, despite these benefits, breastfeeding rates have not yet reached desired levels in many countries today.

The World Health Organization (WHO) and the United Nations Children's Fund (UNICEF) recommend that during the first six months, infants should be exclusively breastfed, avoiding the use of water, other liquids, supplementary foods/formula, and solid foods.In our country, according to the Turkey Demographic and Health Survey 2018 data, the rate of exclusive breastfeeding during the first six months is 41%. Among these mothers, it has been determined that 41.7% of them provide their babies with additional liquids/foods other than breast milk within the first three days after birth. Contrary to recommendations, the use of additional liquids/foods in the early days increases the risk of discontinuing breastfeeding before six months by threefold.

Regardless of medical reasons, the main reasons for the consumption of supplementary foods/formula in the early days include the baby's frequent hunger cues and the mother's concern that her milk might not be sufficient. Additionally, the physiological weight loss that newborns experience in the first few days after birth further supports and amplifies mothers' concerns of "not having enough milk." After the 3rd to 5th day following birth, as milk production advances in the mother's body, the subsequent process involves milk becoming fattier and the baby beginning to gain weight. Therefore, it is crucial for mothers to be properly informed about this process, including the baby's behaviors and the content of the milk.

In addition to these physiological changes, Freud has developed a theory on psychosexual development. At the core of the theory lies a pleasurable pursuit for bodily sensations and control. The period from birth to one year of age is referred to as the "Oral Stage" in that theory. During this period, it is emphasized that the newborn starts to explore the world orally and derives satisfaction/pleasure from sucking behavior. Examples of this are finger sucking, pacifier use, and the behavior of putting any object they hold into their mouth, commonly observed in babies. These are typical processes of a healthy newborn and a developing baby within the context of psychosexual development over time. Hence, infants can exhibit hunger cues not only to satisfy their hunger but also for the purpose of experiencing pleasure. However, no study in the literature has directly correlated this information with newborn-sucking behavior. Current research underscores the need for effective interventions with proper timing and highlights that primiparous mothers tend to have greater concerns about insufficient milk than multiparous mothers. Proper guidance and information about physiological processes are crucial for acquiring breastfeeding behavior. In this study, in line with Freud's psychosexual development theory, the impact of breastfeeding education provided after childbirth on primiparous mothers' feeding attitudes and behaviors has been investigated.

ELIGIBILITY:
Inclusion Criteria:

* being primitive,
* being 18 years or older,
* having a healthy birth,
* using a mobile phone,
* being within 72-96 hours after birth,
* participating in the research voluntarily.

Exclusion Criteria:

* having cognitive problems,
* delivering a premature newborn, having a baby in the neonatal intensive care unit,
* having a health problem that would prevent her from breastfeeding the baby,
* using any sedatives, anticonvulsants, or analgesics, don't the ability to speak Turkish,
* giving formula to their baby for any reason within the first three days,
* having a life-threatening illness or condition,
* not being willing to participate in the study will be excluded.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The study was carried out with mothers who gave birth, so women were studied.
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
IOWA Infant Feeding Attitude Scale | 1 WEEK
  The scale was developed by De La Mora et al. in 1999 to assess the attitudes of women towards breastfeeding and to predict the choice of infant feeding method as well as the duration of breastfeeding. The total attitude score ranges from 17 (indicating a positive attitude towards bottle feeding) to 85 (reflecting a positive attitude towards breastfeeding).
Breastfeeding Form | 1 WEEK
  This form was created by the researchers to evaluate the mothers' experiences of breastfeeding and using formula for one week after birth. The form includes four questions about breastfeeding frequency & duration and formula use & frequency from day to day.

CONTACTS AND LOCATIONS:
Overall Officials: Eyşan Hanzade UMAÇ, Principal Investigator — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Savas EH, Semerci R, Eroglu K, Can N, Ozturk A. Impact of psychosexual development theory-based breastfeeding education on infant feeding attitudes and knowledge of primiparous mothers: A randomized controlled study. J Pediatr Nurs. 2024 Jul-Aug;77:e503-e510. doi: 10.1016/j.pedn.2024.05.016. Epub 2024 May 18. PMID 38762425